CLINICAL TRIAL: NCT01939977
Title: Efficacy and Safety of Paricalcitol in the Reduction of Secondary Hyperparathyroidism After Renal Transplantation.
Brief Title: Efficacy and Safety of Paricalcitol in the Reduction of Secondary Hyperparathyroidism After Kidney Transplantation.
Acronym: PARIDOINAL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fundación Senefro (Other)
Collaborators: AbbVie (Industry); Effice Servicios Para la Investigacion S.L. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACA-SPAI-11-24; 2013-001326-25 (EudraCT Number)
Record Dates: First submitted 2013-08-28; First posted 2013-09-11 (Estimated); Results first posted 2018-11-19 (Actual); Last update posted 2018-11-19 (Actual); Status verified 2018-05

CONDITIONS: Secondary Hyperparathyroidism Due to Renal Causes
Keywords: Hyperparathyroidism; Hyperparathyroidism Secondary; Paricalcitol; Calcifediol; Parathyroid hormone; Renal transplantation
MeSH Terms: conditions — Hyperparathyroidism; Hyperparathyroidism, Secondary | interventions — paricalcitol; Calcifediol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Paricalcitol (Experimental): Paricalcitol oral capsules.
  Interventions: Drug: Paricalcitol
- Calcifediol (Active Comparator): Calcifediol oral drops.
  Interventions: Drug: Calcifediol

INTERVENTIONS:
Drug: Paricalcitol — 1 capsule/day for 6 months. On Month 1 and Month 3 it can be increased up to 2 capsules/day or decreased down to 1 capsule/48 hours.
  Other Names: Zemplar
  Arms: Paricalcitol
Drug: Calcifediol — 5 drops/day during 6 months. On Month 1 it can be increased up to 7 drops/day. If this occurs then, on Month 3, it can decreased to 5 drops/day or continue 7 drops/day until end of treatment.
  Other Names: Hidroferol
  Arms: Calcifediol

SUMMARY:
To demonstrate the superiority of paricalcitol treatment at early renal post-transplantation (M6) in the control of iPTH (Intact parathyroid hormone) compared to the use of vitamin D nutritional supplements (calcifediol) in patients with renal transplantation.

DETAILED DESCRIPTION:
The purpose of this study is to demonstrate the superiority of paricalcitol treatment at early renal post-transplantation (M6) in the control of iPTH (Intact parathyroid hormone) compared to the use of vitamin D nutritional supplements (calcifediol) in patients with renal transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Patient that have willingly signed and dated the ICD (Informed Consent Document) approved by the EC (Ethics Committee) before any study procedure and after they have been explained the study, they have read the ICD and have had the opportunity to make questions about it.
* Patients of both genders and older than 18 years candidates to an immediately renal transplantation from living or deceased donor.
* 24 hours previous to the transplantation, patient must have a significant grade of secondary hyperparathyroidism, defined as iPTH (Intact parathyroid hormone) levels between 110 and 600 pg/mL as per central laboratory results.
* Patients with a preformed antibody panel <20% 24 hours before the transplantation or that are considered by the investigator of low immunological risk (PRA determination is being done on local laboratory, not central).
* Serum calcium (corrected by albumin) < 10 mg/dL 24 hour previous to the transplantation as per central laboratory results.
* Patients that are to be treated with immunosuppression based on tacrolimus, mofetil mycofenolate or mycophenolic acid and with steroids and that are not going to be treated with mTOR (mammalian target of rapamycin) inhibitors. Tacrolimus and steroids must not be removed on the 6 month post-transplantation.
* Patients that are able to take oral capsules on the first week post-transplantation.

Exclusion Criteria:

* Third or subsequent renal transplantation.
* Positive cross-match assay or ABO (A-B-0) incompatibility
* Patients that have been or are going to be recipients of other organs other than the kidney or a double kidney transplantation.
* Patients with history of allergic reaction or sensibility to paricalcitol, calcifediol or similar study drugs (related with vitamin D).
* Patients with chronic gastrointestinal disease, that, based on investigators criteria, can cause significant gastrointestinal malabsorption.
* Patient with hypo or hyperthyroidism not controlled based on investigators criteria.
* Patient with uncontrolled hypertension based on investigators criteria.
* Patients that, 48 hours previous to transplantation, have been receiving calcimimetics.
* Patients with VIH (human immunodeficiency virus)infection of positive serology for HBV (hepatitis B virus) and/or HCV (hepatitis C virus)
* Patients on treatment with drugs contraindicated with paricalcitol and calcifediol (based on SMPC)
* Patients that are participating on other clinical trial with investigational drugs.
* Women of childbearing potential (defined as those whose last menstruation was <2 years ago and that are not surgically sterilized) that are not willing to use correct contraception during study treatment.
* Patient with other diseases or conditions that based on investigators criteria are not suitable for the study.
* Treatment will not be started if the Calcium-Phosphorus product (CAxP)is >55 mg2/dL2 or in case of hyperphosphatemia considered significant as per investigator criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2014-01; Primary Completion 2015-09 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Josep M Cruzado, Dr, Principal Investigator — Fundación SENEFRO - Hospital Universitario de Bellvitge - Barcelona.
Locations (16):
- Spain (16):
  - Hospital Universitari Germans Trias I Pujol de Badalona, Badalona, Barcelona
  - Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario Marqués de Valdecilla, Santander, Cantabria
  - Complexo Hospitalario Universitario A Coruna, A Coruña
  - Hospital Del Mar, Barcelona
  - Fundació Puigvert-Iuna, Barcelona
  - Hospital Universitari Vall D'Hebron, Barcelona
  - Hospital Puerta Del Mar, Cadiz
  - Hospital Reina Sofía, Córdoba
  - Complejo Hospitalario Universitario de Canarias, Las Palmas de Gran Canaria
  - Hospital Ramón Y Cajal, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Complejo Hospitalario Regional de Málaga, Málaga
  - Hospital Virgen Del Rocío, Seville
  - Hospital Universitari I Politècnic La Fe, Valencia
  - Hospital Universitario Miguel Servet, Zaragoza

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 94 patients were randomized, but a total of 148 patients were recruited from January 2014 to February 2015.
Pre-assignment Details: 54 of 148 patients were excluded: 48 due to Screening failure and 6 for other reasons.
Period: Overall Study
Arm/Group | Paricalcitol | Calcifediol
Started | 46 | 48 (48 patients randomized but 1 did not meet inclusion criteria. 47 patients analyzed.)
Completed | 37 | 41
Not Completed | 9 | 7
Not completed — Adverse Event | 4 | 3
Not completed — Lack of Efficacy | 3 | 0
Not completed — Physician Decision | 1 | 1
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Did not meet inclusion criteria | 1 | 0
Not completed — Did not receive study medication | 0 | 1

BASELINE CHARACTERISTICS:
Population: 48 patients were randomized to Calcifediol but 1 patient did not receive study medication because patient did not meet inclusion criteria. So total number of patients that were randomized and started Calcifediol was 47. Total randomized patients: 46+47=93
Groups:
- Total: Total of all reporting groups
Arm/Group | Paricalcitol | Calcifediol | Total
Number analyzed (Participants) | 46 | 47 | 93
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.93 (13.05) | 56.15 (14.48) | 57.53 (13.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 16 | 30
  Male | 32 | 31 | 63

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With iPTH Serum Concentration >110 pg/mL.
Description: Percentage of patients with iPTH serum concentration >110 pg/mL 6 month after transplant.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Paricalcitol | Calcifediol
Number analyzed (Participants) | 46 | 47
Participants
  iPTH>110 pg/ml | 9 | 16
  iPTH<=110 pg/ml | 32 | 27
  N missing | 5 | 4
Statistical Analysis 1: Comparison: Paricalcitol vs Calcifediol; Taking "per protocol" population, the percentage of patients with iPTH> 110 pg / ml at 6 months post-transplant treated with Paricalcitol was statistically lower than in patients treated with Calcifediol; Test type: Superiority; p = 0.0083, Chi-squared

2. Secondary Outcome: Change on iPTH Serum Concentration. Intention to Treat Analysis.
Description: Change on iPTH serum concentration on each treatment group 6 month post transplantation.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: iPTH pg/ml
Arm/Group | Paricalcitol | Calcifediol
Number analyzed (Participants) | 41 | 43
iPTH pg/ml
  iPTH at month 6 | 75.63 (55.5) | 101.27 (55.1)
  iPTH at baseline | 338.48 (135.3) | 315.47 (117.7)

3. Secondary Outcome: Percentage of Patients That Reach at Least a 30% iPTH Reduction at the End of the Study.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Paricalcitol | Calcifediol
Number analyzed (Participants) | 46 | 47
Participants
  Reduction iPTH>=30% | 39 | 38
  Reduction iPTH<30% | 2 | 5
  N missing | 5 | 4

4. Secondary Outcome: Percentage of Patients With iPTH Levels Between 70-110 pg/mL at the End of the Study. ITT.
Time Frame: 6 month
Measure: Count of Participants; unit: Participants
Arm/Group | Paricalcitol | Calcifediol
Number analyzed (Participants) | 41 | 43
Participants
  iPTH<70 pg/ml | 26 | 16
  iPTH 70-110 pg/ml | 6 | 11
  iPTH >110 pg/ml | 9 | 16

5. Secondary Outcome: Percentage of Patient With Presence of Calcifications on Protocol Renal Biopsies at 6 Months After Treatment in Each Treatment Group.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Paricalcitol | Calcifediol
Number analyzed (Participants) | 17 | 19
Participants
  Calcifications | 1 | 0
  No calcifications | 16 | 19

6. Secondary Outcome: Patients That Suffered the Following Events: Acute Rejection, Acute Rejection Confirmed With Biopsy and/or Subclinic Rejection and/or Chronic Damage.
Description: Patients with at least one of the following events: acute rejection, acute rejection confirmed with biopsy and/or subclinic rejection and/or chronic damage.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Paricalcitol | Calcifediol
Number analyzed (Participants) | 46 | 47
Participants
  Patients with at least one event | 14 | 6
  Patients with no events | 12 | 15
  N missing | 20 | 26

7. Secondary Outcome: Change on Concentration of Bone Markers (Osteocalcin) at 6 Months After Transplantation on Each Treatment Group.
Time Frame: 6 months
Population: This value was missing for some patients at month 6
Measure: Mean (Standard Deviation); unit: Osteocalcin ng/ml
Arm/Group | Paricalcitol | Calcifediol
Number analyzed (Participants) | 46 | 47
Osteocalcin ng/ml
  Baseline Osteocalcin | 11.74 (9.2) | 12.62 (8.5)
  Month 6 Osteocalcin: number analyzed (Participants) | 42 | 41
  Month 6 Osteocalcin | 4.02 (3.6) | 5.20 (4.1)

8. Secondary Outcome: Percentage of Patients With Acute Rejection at 6 Months After Transplantation and Treatment on Each Treatment Group.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Paricalcitol | Calcifediol
Number analyzed (Participants) | 46 | 47
Participants
  Yes | 5 | 2
  No | 41 | 45

9. Secondary Outcome: Percentage of Patients With Microalbuminuria on Months 1, 3 and 6 Post Transplantation.
Time Frame: Months 1, 3 and 6
Measure: Count of Participants; unit: Participants
Arm/Group | Paricalcitol | Calcifediol
Number analyzed (Participants) | 46 | 47
Participants
  Microalbuminuria month 1: Normal (UACR<30 mg/g) | 18 | 16
  Microalbuminuria month 1: UACR 30-300 mg/g | 3 | 1
  Microalbuminuria month 1: N missing | 25 | 30
  Microalbuminuria month 3: Normal (UACR<30 mg/g) | 13 | 12
  Microalbuminuria month 3: UACR 30-300 mg/g | 3 | 0
  Microalbuminuria month 3: N missing | 30 | 35
  MIcroalbuminuria month 6: Normal (UACR<30 mg/g) | 16 | 14
  MIcroalbuminuria month 6: UACR 30-300 mg/g | 1 | 0
  MIcroalbuminuria month 6: N missing | 29 | 33

10. Secondary Outcome: Percentage of Patients on Each Stage of Renal Function on Months 1, 3 and 6 Post Transplantation.
Time Frame: Months 1, 3 and 6
Measure: Count of Participants; unit: Participants
Arm/Group | Paricalcitol | Calcifediol
Number analyzed (Participants) | 46 | 47
Participants
  Renal function at month 1: eGFR >=90 | 1 | 4
  Renal function at month 1: eGFR 60-89 | 5 | 5
  Renal function at month 1: eGFR 30-59 | 29 | 27
  Renal function at month 1: eGFR 15-29 | 6 | 9
  Renal function at month 1: eGFR<15 | 3 | 1
  Renal function at month 1: N missing | 2 | 1
  Renal function at month 3: eGFR >=90 | 2 | 2
  Renal function at month 3: eGFR 60-89 | 2 | 10
  Renal function at month 3: eGFR 30-59 | 26 | 25
  Renal function at month 3: eGFR 15-29 | 8 | 8
  Renal function at month 3: eGFR<15 | 2 | 0
  Renal function at month 3: N missing | 6 | 2
  Renal function at month 6: eGFR >=90 | 1 | 3
  Renal function at month 6: eGFR 60-89 | 5 | 9
  Renal function at month 6: eGFR 30-59 | 24 | 25
  Renal function at month 6: eGFR 15-29 | 9 | 5
  Renal function at month 6: eGFR<15 | 2 | 1
  Renal function at month 6: N missing | 5 | 4

11. Secondary Outcome: Evolution of Speed of Pulse Wave From Month 1 to Month 6 Post Transplantation.
Description: Baseline speed of pulse wave was performed between 1 week and 1 month post transplant; next measure of speed of pulse wave performed at month 6 post transplant.
Time Frame: 6 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Paricalcitol | Calcifediol
Number analyzed (Participants) | 17 | 14
Participants
  Speed pulse wave gets better at month 6 | 1 | 1
  Speed pulse wave maintained | 14 | 12
  Speed pulse wave gets worse at month 6 | 2 | 1

12. Secondary Outcome: Percentage of Patients With Hypercalcemia on Each Treatment Group at 6 Months Post Transplantation.
Description: Percentage of patients with hypercalcemia (defined as serum calcium levels > 10,3 mg/dl) on each treatment group at 6 months post transplantation.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Paricalcitol | Calcifediol
Number analyzed (Participants) | 46 | 47
Participants
  Serum Ca >10,3 mg/dl | 3 | 2
  Serum Ca <=10,3 mg/dl | 39 | 41
  N missing | 4 | 4

13. Secondary Outcome: Evolution of Anti-HLA Antibodies (PRA) From Basal to Month 6 Post-transplantation.
Description: HLAs corresponding to MHC (major histocompatibility complex) class I (A, B, and C) present peptides from inside the cell. HLAs corresponding to MHC class II (DP, DM, DO, DQ, and DR) present antigens from outside of the cell to T-lymphocytes.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Paricalcitol | Calcifediol
Number analyzed (Participants) | 40 | 42
Participants
  Screening Luminex at transplant: Positive class I | 1 | 0
  Screening Luminex at transplant: Positive class II | 3 | 4
  Screening Luminex at transplant: Positive class I and II | 1 | 1
  Screening Luminex at transplant: Negative | 35 | 37
  Screening Luminex at month 6: Positive class I | 1 | 0
  Screening Luminex at month 6: Positive class II | 6 | 3
  Screening Luminex at month 6: Positive class I and II | 1 | 1
  Screening Luminex at month 6: Negative | 32 | 38

14. Secondary Outcome: Frequency of Adverse Events or Serious Adverse Events That Occurs During the Study on Each Treatment Group.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Paricalcitol | Calcifediol
Number analyzed (Participants) | 46 | 47
Participants
  Patients with adverse event (AE) | 41 | 38
  Patients with possibly or probably related AE | 2 | 1
  Patients with serious adverse event (SAE) | 24 | 20
  Patients with possibly or probably related SAE | 0 | 0
  Patients with AE that leads to discontinuation | 2 | 4
  Patients with moderate-severe adverse event | 34 | 28

15. Secondary Outcome: Change on Concentration of Bone Markers (Alkaline Phosphatase) at 6 Months After Transplantation on Each Treatment Group.
Time Frame: 6 months
Population: This value was missing for some patients at month 6
Measure: Mean (Standard Deviation); unit: ug/L
Arm/Group | Paricalcitol | Calcifediol
Number analyzed (Participants) | 46 | 47
ug/L
  Baseline alkaline phosphatase | 13.85 (6.9) | 14.50 (7.4)
  Month 6 alkaline phosphatase: number analyzed (Participants) | 42 | 42
  Month 6 alkaline phosphatase | 11.68 (9.1) | 11.79 (5.1)

16. Secondary Outcome: Change on Concentration of Bone Markers (FGF-23) at 6 Months After Transplantation on Each Treatment Group
Time Frame: 6 months
Population: This value was missing for some patients
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Paricalcitol | Calcifediol
Number analyzed (Participants) | 46 | 47
pg/mL
  Baseline FGF-23 | 2039.13 (3559.8) | 1359.56 (7112.9)
  Month 6 FGF-23: number analyzed (Participants) | 42 | 42
  Month 6 FGF-23 | 1937.30 (3738.0) | 289.14 (945.1)

ADVERSE EVENTS:
Time Frame: Adverse events collected during the participation in the study (6 months). Non serious adverse events: only reported here the study medication related adverse events.
Arm/Group | Paricalcitol | Calcifediol
All-Cause Mortality (participants affected / at risk) | 0/46 | 0/47
Serious Adverse Events (participants affected / at risk) | 24/46 | 20/47
Other Adverse Events (participants affected / at risk) | 2/46 | 1/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Paricalcitol (N=46) | Calcifediol (N=47)
Infections (Infections and infestations) | 11 (11) | 6 (7)
Surgical wound (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Transitional cells carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Transplantectomy (Surgical and medical procedures) | 0 | 1
Lymphocele marsupialization (Surgical and medical procedures) | 1 | 0
Heart failure (Cardiac disorders) | 1 (1) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Impaired renal function (Renal and urinary disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Allograft rejection (Immune system disorders) | 1 (1) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Metabolic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Anal bleeding (Gastrointestinal disorders) | 0 (0) | 1 (1)
Extravasation (General disorders) | 0 (0) | 1 (1)
Pirexia (General disorders) | 2 (2) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Acute cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Positive test for Pseudomonas (Infections and infestations) | 0 (0) | 1 (1)
Impaired renal function (Renal and urinary disorders) | 7 (8) | 3 (3)
Ureteral dilation (Renal and urinary disorders) | 1 (1) | 0 (0)
Hematuria (Renal and urinary disorders) | 0 (0) | 2 (2)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Hyperpotasemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Dehydratation (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Acute pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hematoma (Vascular disorders) | 0 (0) | 1 (1)
Lymphocele (Vascular disorders) | 1 (2) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Paricalcitol (N=46) | Calcifediol (N=47)
Parotiditis (Endocrine disorders) | 0 (0) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No